CLINICAL TRIAL: NCT02370615
Title: A Phase 1, Drug-Drug Interaction Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of TAK-272 and the Effect of TAK-272 on the Pharmacokinetics of Digoxin or Midazolam In the Healthy Adult Participants
Brief Title: Drug-Drug Interaction Study Between TAK-272 and Itraconazole, Digoxin or Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-272/CPH-011; U1111-1167-0017 (Registry Identifier: WHO); JapicCTI-152810 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Japanese Healthy Adult Males
MeSH Terms: interventions — imarikiren hydrochloride; Digoxin; Itraconazole; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: TAK-272 + Itraconazole (Experimental): TAK-272 40 mg, tablet, orally, once on Day 1 and 10, followed by Itraconazole 200 mg, solution, orally, twice on Day 4, further followed by Itraconazole 200 mg, solution, orally, once from Day 5 to 12.
  Interventions: Drug: TAK-272; Drug: Itraconazole
- Cohort 2: Midazolam + Digoxin + TAK-272 (Experimental): Midazolam 2 mg, syrup, and Digoxin 0.25 mg, tablet, orally, once on Day 1 and 7, followed by TAK-272 80 mg, tablet, orally, once from Day 3 to 8.
  Interventions: Drug: TAK-272; Drug: Digoxin; Drug: Midazolam

INTERVENTIONS:
Drug: TAK-272 — TAK-272 tablet.
Drug: Digoxin — Digoxin tablet.
  Arms: Cohort 2: Midazolam + Digoxin + TAK-272
Drug: Itraconazole — Itraconazole oral solution
  Arms: Cohort 1: TAK-272 + Itraconazole
Drug: Midazolam — Midazolam syrup.
  Arms: Cohort 2: Midazolam + Digoxin + TAK-272

SUMMARY:
The purpose of this study is to evaluate the effect of repeated-dose administration of itraconazole on the pharmacokinetics of TAK-272, as well as the effect of repeated-dose administration of TAK-272 on the pharmacokinetics of digoxin or midazolam in healthy Japanese adult males.

DETAILED DESCRIPTION:
In Cohort 1, the effect of repeated-dose administration of itraconazole on the pharmacokinetics of TAK-272 was evaluated by comparing between participants receiving TAK-272 alone and those receiving TAK-272 in combination with itraconazole. In Cohort 2, the effect of repeated-dose administration of TAK-272 on the pharmacokinetics of digoxin or midazolam was evaluated by comparing between participants receiving digoxin or midazolam alone and those receiving either of the drugs in combination with TAK-272.

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding and complying with protocol requirements.
2. Who can sign and date the informed consent form before the initiation of the study procedure.
3. Healthy Japanese adult male volunteer.
4. Is of 20 to 35 years of age at the time of informed consent
5. Weighs 50 kilogram (kg) or more with a body mass index (BMI) of 18.5 to less than 25.0 kilogram per square meter (kg/m^2) at the screening test.
6. Male participant who was nonsterilized and sexually active with a female partner of childbearing potential had to agree to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after the completion of the study.

Exclusion Criteria:

1. Who was administered any investigational product within 16 weeks (112 days) prior to the initial drug administration.
2. Who has received TAK-272 in previous.
3. Employees of the study site, their family members, those who are in a dependency relationship with employees of the study site involved in the conduct of the study (example, spouse, parents, children, brothers and sisters), or those who might be coerced to consent to participate in the study.
4. Who has poorly controlled, clinically significant abnormalities of the nervous system, cardiovascular system, lungs, liver, kidneys, metabolism, gastrointestinal system, urinary system, endocrinological system or other organs or systems, and which may possibly affect study participation or study results.
5. Who has a history of serious hepatic disease.
6. Who has atrioventricular block or sinoatrial block.
7. Has digitalis intoxication.
8. Has acute narrow-angle glaucoma.
9. Has myasthenia gravis.
10. Has hypersensitivity to TAK-272 or any other renin inhibitors.
11. Has hypersensitivity to itraconazole, digoxin, digitalis preparation, or midazolam.
12. Has allergy to cherries.
13. Has a positive to urine test for drug abuse at the screening.
14. Has a history of drug abuse (defined as illegal drug use) or alcohol addiction within 1 year prior to the screening visit, and those who are not willing to give up alcohol or drugs during the study period.
15. Who needs to use prohibited concomitant drugs, vitamins, or foods listed in the table of prohibited concomitant drugs and foods, and the participant who has used any of them during the period prohibiting the concomitant use.
16. Male participants who plans to donate sperm during the study period or up to 12 weeks after the end of the study.
17. Who currently has cardiovascular, central nervous, hepatic, or hematopoietic disease, renal insufficiency, metabolic or endocrinological disorder, serious allergy, asthma, hypoxemia, hypertension, convulsions, or allergic rash.
18. Has a disease history, examination findings, or clinical test findings related to safety that reasonably suggest a disease for which TAK 272 or related renin inhibitors in the same class, itraconazole, digoxin, or midazolam is contraindicated or a disease that may affect the study conduct (which includes, for example, peptic ulcer disease, convulsive disorder, and arrhythmia).
19. Who currently has or recently had (within the past 6 months) gastrointestinal disease that may affect drug absorption (malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [at least once a week] heartburn, surgical intervension [e.g., cholecystectomy]).
20. Has past history of cancer.
21. Who is positive for any of the following at screening: hepatitis B virus surface antigen (HBs), antibody against hepatitis C virus (HCV), human immunodeficiency virus (HIV) antigen, anti-HIV antibody, or serological tests for syphilis.
22. The participant with difficulty having blood collected from a peripheral vein.
23. Who has donated 200 milliliter (mL) or more whole blood within the 4 weeks (28 days) or 400 mL or more whole blood within the 12 weeks (84 days) before starting the study drug administration.
24. Who has donated a total of 800 mL or more of whole blood within the 52 weeks (364 days) before the day of starting the study drug administration.
25. Who has donated blood components within the 2 weeks (14 days) before starting the study drug administration.
26. Who shows clinically significant abnormalities in electrocardiogram at screening or before the study drug administration.
27. Who shows laboratory test abnormalities suggestive of a clinically significant primary disease or who shows abnormal values in any of the following parameters at screening or before the study drug administration: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) exceeding 1.5 times the upper limit of the normal range.
28. Who is unlikely to comply with the study protocol or is ineligible for the study for any other reason, as considered by the investigator or sub investigator.
29. Who had systolic blood pressure under 80 millimeter of mercury(mmHg) at Screening, pretreatment examination, and before the start of study drug administration, and who had suspected hypotension with 2 or more of the following symptoms and findings through physical examinations: dizziness postural, facial pallor, cold sweat.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda
Locations (1):
- Osaka, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 25-February-2015 to 16-April-2015.
Pre-assignment Details: Healthy Japanese adult male participants were enrolled to receive TAK-272 and itraconazole in cohort 1 or TAK-272 and digoxin/midazolam in cohort 2.
Groups:
- Cohort 1: TAK-272 + Itraconazole: TAK-272 40 milligram (mg), tablet, orally, once on Day 1 and 10, followed by Itraconazole 200 mg, solution, orally, twice on Day 4, further followed by Itraconazole 200 mg, solution, orally, once from Day 5 to 12.
Period: Overall Study
Arm/Group | Cohort 1: TAK-272 + Itraconazole | Cohort 2: Midazolam + Digoxin + TAK-272
Started | 16 | 18
Completed | 15 | 18
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic analysis set was defined as the set of participants treated with the study drug that had no significant protocol deviation, satisfied the minimum protocol provisions, and could be evaluated for pharmacokinetics.
Groups:
- Cohort 2: Midazolam + Digoxin + TAK-272: Midazolam 2 mg, syrup, and Digoxin 0.25 mg, tablet, orally, once on Day 1 and 7, followed by TAK-272 80 mg, tablet, orally, once on Day 3 to 8.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: TAK-272 + Itraconazole | Cohort 2: Midazolam + Digoxin + TAK-272 | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (4.11) | 25.3 (4.44) | 26.0 (4.30)
Sex/Gender, Customized [Number; unit: participants]
  Male | 15 | 18 | 33
Smoking Classification [Number; unit: participants]
  Never smoked | 12 | 12 | 24
  Current smoker | 1 | 1 | 2
  Ex-smoker | 2 | 5 | 7
Alcohol Classification [Number; unit: participants]
  Drinks a few days per week | 5 | 2 | 7
  Drinks a few days per month | 5 | 5 | 10
  Does not drink | 5 | 11 | 16
Caffeine Classification [Number; unit: participants]
  Caffeine consumption | 7 | 6 | 13
  No caffeine consumption | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK 272F and TAK 272-Metabolite (M-I) in Cohort 1
Time Frame: Day 1 and Day 10: pre-dose and at multiple time-points (upto 72 hours) postdose; Day 1 for Cohort 1: TAK-272 and Day 10 for Cohort 1: TAK-272 + Itraconazole
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Cohort 1: TAK-272: TAK-272 40 mg, tablet, orally, once on Day 1.
- Cohort 1: TAK-272 + Itraconazole: TAK-272 40 mg, tablet, orally, once on Day 10, followed by Itraconazole 200 mg, solution, orally, twice on Day 4, further followed by Itraconazole 200 mg, solution, orally, once from Day 5 to 12.
Arm/Group | Cohort 1: TAK-272 | Cohort 1: TAK-272 + Itraconazole
Number analyzed (Participants) | 15 | 15
nanogram per milliliter (ng/mL)
  TAK 272 | 387.8 (286.18) | 780.3 (258.45)
  TAK 272-M-I | 10.02 (7.1545) | 0.9550 (0.55302)
Statistical Analysis 1: Comparison: Cohort 1: TAK-272 vs Cohort 1: TAK-272 + Itraconazole; Analysis for TAK 272F; Test type: Superiority or Other; Geometric Mean Ratio (Day 10/Day 1) = 2.012, 90% CI 2-sided [1.632 to 2.481]
Statistical Analysis 2: Comparison: Cohort 1: TAK-272 vs Cohort 1: TAK-272 + Itraconazole; Analysis for TAK 272-M-I; Test type: Superiority or Other; Geometric Mean Ratio (Day 10/Day 1) = 0.089, 90% CI 2-sided [0.064 to 0.123]

2. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK 272F and TAK 272-M-I in Cohort 1
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | Cohort 1: TAK-272 | Cohort 1: TAK-272 + Itraconazole
Number analyzed (Participants) | 15 | 15
nanogram hours per milliliter (ng*hr/mL)
  TAK 272 | 1861 (731.14) | 9098 (2809.8)
  TAK 272-M-I | 46.53 (19.347) | 9.373 (8.9682)
Statistical Analysis 1: Comparison: Cohort 1: TAK-272 vs Cohort 1: TAK-272 + Itraconazole; Analysis for TAK 272F; Test type: Superiority or Other; Geometric Mean Ratio (Day 10/Day 1) = 4.888, 90% CI 2-sided [4.137 to 5.777]

3. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK 272F and TAK 272-M-I in Cohort 1
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-272 | Cohort 1: TAK-272 + Itraconazole
Number analyzed (Participants) | 15 | 15
ng*hr/mL
  TAK 272 | 1842 (728.15) | 8659 (2596.7)
  TAK 272-M-I | 38.34 (16.944) | 0.9092 (1.5900)
Statistical Analysis 1: Comparison: Cohort 1: TAK-272 vs Cohort 1: TAK-272 + Itraconazole; Analysis for TAK 272F; Test type: Superiority or Other; Geometric Mean Ratio (Day 10/Day 1) = 4.702, 90% CI 2-sided [3.969 to 5.569]
Statistical Analysis 2: Comparison: Cohort 1: TAK-272 vs Cohort 1: TAK-272 + Itraconazole; Analysis for TAK 272-M-I; Test type: Superiority or Other; Geometric Mean Ratio (Day 10/Day 1) = 0.023, 90% CI 2-sided [0.012 to 0.045]

4. Primary Outcome: Cumulative Urinary Excretion Ratio of TAK 272F and TAK 272-M-I From 0 to 72 Hours Postdose in Cohort 1
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Cohort 1: TAK-272 | Cohort 1: TAK-272 + Itraconazole
Number analyzed (Participants) | 15 | 15
percentage of dose
  TAK 272 | 11.523 (2.6615) | 37.803 (5.4878)
  TAK 272-M-I | 0.556 (0.1534) | 0.071 (0.0467)

5. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Digoxin in Cohort 2
Time Frame: Day 1 and Day 7: pre-dose and at multiple time-points (upto 48 hours) postdose; Day 1 for Cohort 2: Digoxin and Day 7 for Cohort 2: Digoxin + TAK-272
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 2: Digoxin: Digoxin 0.25 mg, tablet, orally once on Day 1 and 7.
- Cohort 2: Digoxin + TAK-272: Digoxin 0.25 mg, tablet, orally once on Day 7, further followed by TAK-272 80 mg, tablet, orally, once from Day 3 to 8.
Arm/Group | Cohort 2: Digoxin | Cohort 2: Digoxin + TAK-272
Number analyzed (Participants) | 18 | 18
ng/mL | 1.212 (0.58104) | 1.635 (0.70089)
Statistical Analysis 1: Comparison: Cohort 2: Digoxin vs Cohort 2: Digoxin + TAK-272; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 1.349, 90% CI 2-sided [1.117 to 1.628]

6. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Digoxin in Cohort 2
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 2: Digoxin | Cohort 2: Digoxin + TAK-272
Number analyzed (Participants) | 18 | 18
ng*hr/mL | 15.49 (4.4007) | 15.79 (4.2495)
Statistical Analysis 1: Comparison: Cohort 2: Digoxin vs Cohort 2: Digoxin + TAK-272; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 1.020, 90% CI 2-sided [0.919 to 1.131]

7. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Digoxin in Cohort 2
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 2: Digoxin | Cohort 2: Digoxin + TAK-272
Number analyzed (Participants) | 18 | 18
ng*hr/mL | 9.191 (2.6150) | 10.61 (2.6705)
Statistical Analysis 1: Comparison: Cohort 2: Digoxin vs Cohort 2: Digoxin + TAK-272; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 1.155, 90% CI 2-sided [1.035 to 1.289]

8. Primary Outcome: Urinary Excretion Ratio of Digoxin From 0 to 48 Hours Postdose in Cohort 2
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Cohort 2: Digoxin | Cohort 2: Digoxin + TAK-272
Number analyzed (Participants) | 18 | 18
percentage of dose | 31.391 (8.4376) | 35.983 (7.7691)

9. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Midazolam and 1'Hydroxymidazolam in Cohort 2
Time Frame: Day 1 and Day 7: pre-dose and at multiple time-points (upto 24 hours) postdose; Day 1 for Cohort 2: Midazolam and Day 7 for Cohort 2: Midazolam + TAK-272
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 2: Midazolam: Midazolam 2 mg, syrup, orally, once on Day 1.
- Cohort 2: Midazolam + TAK-272: Midazolam 2 mg, syrup, orally, once on Day 7, followed by TAK-272 80 mg, tablet, orally, once from Day 3 to 8.
Arm/Group | Cohort 2: Midazolam | Cohort 2: Midazolam + TAK-272
Number analyzed (Participants) | 18 | 18
ng/mL
  Midazolam | 10.02 (3.6198) | 12.37 (5.0127)
  1'hydroxymidazolam | 4.813 (1.8090) | 4.270 (1.1195)
Statistical Analysis 1: Comparison: Cohort 2: Midazolam vs Cohort 2: Midazolam + TAK-272; Analysis for Midazolam; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 1.235, 90% CI 2-sided [1.100 to 1.387]
Statistical Analysis 2: Comparison: Cohort 2: Midazolam vs Cohort 2: Midazolam + TAK-272; Analysis for 1'Hydroxymidazolam; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 0.887, 90% CI 2-sided [0.781 to 1.008]

10. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Midazolam and 1'Hydroxymidazolam in Cohort 2
Time Frame: as for outcome 9
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 2: Midazolam | Cohort 2: Midazolam + TAK-272
Number analyzed (Participants) | 18 | 18
ng*hr/mL
  Midazolam | 27.11 (11.362) | 38.55 (18.588)
  1'hydroxymidazolam | 13.00 (4.0705) | 14.06 (4.5131)
Statistical Analysis 1: Comparison: Cohort 2: Midazolam vs Cohort 2: Midazolam + TAK-272; Analysis for Midazolam; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 1.422, 90% CI 2-sided [1.290 to 1.568]
Statistical Analysis 2: Comparison: Cohort 2: Midazolam vs Cohort 2: Midazolam + TAK-272; Analysis for 1'Hydroxymidazolam; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 1.081, 90% CI 2-sided [1.008 to 1.160]

11. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Midazolam and 1'Hydroxymidazolam in Cohort 2
Time Frame: as for outcome 9
Population: as for baseline characteristics
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 2: Midazolam | Cohort 2: Midazolam + TAK-272
Number analyzed (Participants) | 18 | 18
ng*hr/mL
  Midazolam | 26.77 (11.343) | 38.16 (18.205)
  1'hydroxymidazolam | 12.49 (3.7079) | 13.25 (3.3695)
Statistical Analysis 1: Comparison: Cohort 2: Midazolam vs Cohort 2: Midazolam + TAK-272; Analysis for Midazolam; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 1.425, 90% CI 2-sided [1.291 to 1.574]
Statistical Analysis 2: Comparison: Cohort 2: Midazolam vs Cohort 2: Midazolam + TAK-272; Analysis for 1'Hydroxymidazolam; Test type: Superiority or Other; Geometric Mean Ratio (Day 7/Day 1) = 1.061, 90% CI 2-sided [0.986 to 1.143]

12. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Cohort 1: Baseline up to Day 19; Cohort 2: Baseline up to Day 15
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Cohort 2: Midazolam + Digoxin + TAK-272: Midazolam 2 mg, syrup, orally, once on Day 1 and 7, followed by Digoxin 0.25 mg, tablet, orally once on Day 1 and 7, further followed by TAK-272 80 mg, tablet, orally, once from Day 3 to 8.
Arm/Group | Cohort 1: TAK-272 + Itraconazole | Cohort 2: Midazolam + Digoxin + TAK-272
Number analyzed (Participants) | 16 | 18
participants | 10 | 7

13. Primary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Cohort 1: Baseline up to Day 19; Cohort 2: Baseline up to Day 15
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: TAK-272 + Itraconazole | Cohort 2: Midazolam + Digoxin + TAK-272
Number analyzed (Participants) | 16 | 18
participants
  Blood pressure decreased | 1 | 0
  Hypotension | 2 | 0
  Heart rate increased | 0 | 1

14. Primary Outcome: Number of Participants With TEAEs Related to Body Weight
Time Frame: Cohort 1: Baseline up to Day 19; Cohort 2: Baseline up to Day 15
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: TAK-272 + Itraconazole | Cohort 2: Midazolam + Digoxin + TAK-272
Number analyzed (Participants) | 16 | 18
participants | 0 | 0

15. Primary Outcome: Number of Participants Who Had Clinically Significant Changes From Baseline in 12-lead Electrocardiograms
Description: Number of participants who had ECG findings changed from "within normal limit" or "abnormal, clinically significant" to "abnormal and clinically significant" after study drug administration.
Time Frame: Cohort 1: Baseline up to Day 19; Cohort 2: Baseline up to Day 15
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: TAK-272 + Itraconazole | Cohort 2: Midazolam + Digoxin + TAK-272
Number analyzed (Participants) | 16 | 18
participants | 0 | 0

16. Primary Outcome: Number of Participants With TEAEs Categorized Into Investigations System Organ Class (SOC) Related to Chemistry, Hematology or Urinalysis
Time Frame: Cohort 1: Baseline up to Day 19; Cohort 2: Baseline up to Day 15
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: TAK-272 + Itraconazole | Cohort 2: Midazolam + Digoxin + TAK-272
Number analyzed (Participants) | 16 | 18
participants
  Alanine aminotransferase increased | 2 | 1
  Blood creatine phosphokinase increased | 1 | 0
  Blood triglycerides increased | 0 | 1
  Urine ketone body present | 0 | 1

17. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Continuous Pulse Oximetry (SpO2) in Cohort 2
Time Frame: Cohort 2: Baseline up to Day 15
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 2: Midazolam + Digoxin + TAK-272
Number analyzed (Participants) | 18
participants | 0

ADVERSE EVENTS:
Time Frame: Collection of AEs commenced from the time that the participant was first administered study drug (Day 1) until the follow-up examination (Day 19 for Cohort 1, Day 15 for Cohort 2)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1: TAK-272 + Itraconazole | Cohort 2: Midazolam + Digoxin + TAK-272
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 10/16 | 7/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: TAK-272 + Itraconazole (N=16) | Cohort 2: Midazolam + Digoxin + TAK-272 (N=18)
Nasopharyngitis (Infections and infestations) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Urine ketone body present (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Dizziness postural (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.